CLINICAL TRIAL: NCT04770285
Title: A Multi-center, Randomized, Controlled Trial to Evaluate the Effectiveness of a Digital Therapeutic (CT-152) as Adjunctive Therapy in Adult Subjects Diagnosed With Major Depressive Disorder
Brief Title: Trial to Evaluate the Effectiveness of a Digital Therapeutics in Adults Diagnosed With Major Depressive Disorder
Acronym: MIRAI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: Click Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 345-201-00002
Record Dates: First submitted 2021-02-19; First posted 2021-02-25 (Actual); Results first posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-09

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Digital Therapeutic A - CT-152 (Other): Participants received digital treatment session by using the CT-152 mobile application (app) from Day 1 up to Week 6 of the treatment period. Each treatment session consisted of Emotional Faces Memory Task (EFMT) exercises and a psychotherapy lesson. From Week 7 up to Week 10 participants continued using the CT-152 app with optional psychotherapy lesson but did not receive any new EFMT exercises during this period. Participants continued receiving brief SMS messages during Weeks 7 to 10 as a reminder of the previously completed CT-152 treatment courses.
  Interventions: Device: CT-152 - Digital Therapeutic
- Digital Therapeutic B - Sham (Other): Participants received digital treatment session by using a sham mobile app from Day 1 up to Week 6 of the treatment period. Each treatment session consisted of a Shape and Memory Task (SMT) exercise only. From Week 7 up to Week 10 participants continued using the sham app but did not receive any new SMT exercises during this period. Participants continued receiving brief SMS messages during Weeks 7 to 10 as a reminder of the previously completed sham treatment courses.
  Interventions: Device: Sham

INTERVENTIONS:
Device: CT-152 - Digital Therapeutic — CT-152 mobile app was used by the participants as per the schedule specified in the respective arm.
  Arms: Digital Therapeutic A - CT-152
Device: Sham — Sham mobile app was used by the participants as per the schedule specified in the respective arm.
  Arms: Digital Therapeutic B - Sham

SUMMARY:
This study compares the effectiveness of 2 digital therapeutics in adult participants diagnosed with major depressive disorder (MDD) who are on antidepressant therapy (ADT) monotherapy for the treatment of depression.

DETAILED DESCRIPTION:
This is a pivotal, 13-week, multi-center, randomized, controlled trial to evaluate the effectiveness and safety of two digital therapeutics in adult participants diagnosed with MDD who are on antidepressant therapy (ADT) monotherapy for the treatment of depression.

The trial consists of a 3-week screening period, a 6-week treatment period, and a 4-week extension. Trial visits will be conducted remotely either by video visit or telephone. The screening visit may be performed in person at the discretion of the investigator. Eligible participants will be randomized to 1 of 2 digital therapeutics within a mobile application that will reside on the participant's personal iPhone or smartphone.

The trial population will include male and female participants between 22 and 64 years of age with a primary diagnosis of major depressive disorder (MDD) who are on an ADT for the treatment of depression. This trial will analyze data gathered from approximately 360 participants in the United States. An interim analysis will be conducted when a targeted sample of the first 180 participants has completed week 6 or discontinued the trial prior to week 6.

ELIGIBILITY:
Key Inclusion Criteria:

* Participants with a current primary diagnosis of MDD.
* Participants with a Hamilton Rating Scale for Depression, 17-item (HAM-D17) score ≥ 18
* Participants who are receiving treatment with an adequate dose and duration of an ADT and who are willing to maintain that same treatment regimen for the duration of this trial.
* Participants who are the only users of an iPhone or an Android smartphone, and agree to download and use the digital mobile application as required by the protocol.

Key Exclusion Criteria:

* Participants with an inadequate response to > 1 adequate trial of ADT for the current episode.
* Participants who are receiving or have received psychotherapy within 90 days prior to screening.
* Participants who are currently using a computer, web, or smartphone software-based application for mental health or depression.
* Participants with a history of schizophrenia, schizoaffective disorder, other psychotic disorder, or Bipolar I/II disorder, or current posttraumatic stress disorder, panic disorder, obsessive-compulsive disorder, or personality disorder
* General Anxiety Disorder/social anxiety can be present as long as they are not the main disorder requiring treatment.

Ages: 22 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 386 (Actual)
Dates: Start 2021-02-25 (Actual); Primary Completion 2022-10-26 (Actual); Study Completion 2022-10-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- For additional information regarding sites, contact 844-687-8522, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on the Vivli data sharing platform which can be found here: https://vivli.org/ourmember/Otsuka/
URL: https://clinical-trials.otsuka.com

REFERENCES:
- [Derived] Rothman B, Slomkowski M, Speier A, Rush AJ, Trivedi MH, Lawson E, Fahmy M, Carpenter D, Chen D, Forbes A. Evaluating the Efficacy of a Digital Therapeutic (CT-152) as an Adjunct to Antidepressant Treatment in Adults With Major Depressive Disorder: Protocol for the MIRAI Remote Study. JMIR Res Protoc. 2024 Aug 20;13:e56960. doi: 10.2196/56960. PMID 39163592

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 37 investigative sites in the United States from 25 February 2021 to 26 October 2022.
Pre-assignment Details: Participants with major depressive disorder were enrolled and randomized in a 1:1 ratio to 1 of the 2 digital mobile applications (CT-152 or sham) on Day 1.
Period: Overall Study
Arm/Group | Digital Therapeutic A - CT-152 | Digital Therapeutic B - Sham
Started | 194 | 192
Full Analysis Set (FAS) (FAS included all randomized participants who received at least 1 occurrence of either CT-152 or sham use and had baseline and at least 1 postbaseline assessment of Montgomery-Asberg Depression Rating Scale (MADRS) total score.) | 177 | 177
Completed | 165 | 164
Not Completed | 29 | 28
Not completed — Non-Compliance With Study Treatment | 3 | 3
Not completed — Lack of Efficacy | 0 | 1
Not completed — Lost to Follow-up | 11 | 8
Not completed — Protocol Deviation | 6 | 6
Not completed — Technical Problem | 0 | 1
Not completed — Withdrawal by Subject | 9 | 8
Not completed — Reason Not Specified | 0 | 1

BASELINE CHARACTERISTICS:
Population: Randomized sample included all participants allocated based on the randomization process and recorded in the database.
Groups:
- Digital Therapeutic A - CT-152: Participants received digital treatment session by using the CT-152 mobile app from Day 1 up to Week 6 of the treatment period. Each treatment session consisted of EFMT exercises and a psychotherapy lesson. From Week 7 up to Week 10 participants continued using the CT-152 app with optional psychotherapy lesson but did not receive any new EFMT exercises during this period. Participants continued receiving brief SMS messages during Weeks 7 to 10 as a reminder of the previously completed CT-152 treatment courses.
- Digital Therapeutic B - Sham: Participants received digital treatment session by using a sham mobile app from Day 1 up to Week 6 of the treatment period. Each treatment session consisted of a SMT exercise only. From Week 7 up to Week 10 participants continued using the sham app but did not receive any new SMT exercises during this period. Participants continued receiving brief SMS messages during Weeks 7 to 10 as a reminder of the previously completed sham treatment courses.
- Total: Total of all reporting groups
Arm/Group | Digital Therapeutic A - CT-152 | Digital Therapeutic B - Sham | Total
Number analyzed (Participants) | 194 | 192 | 386
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.0 (12.1) | 42.2 (12.1) | 42.6 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 165 | 167 | 332
  Male | 29 | 25 | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 16 | 36
  Not Hispanic or Latino | 173 | 174 | 347
  Unknown or Not Reported | 1 | 2 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 141 | 160 | 301
  Black or African American | 36 | 25 | 61
  American Indian or Alaska Native | 5 | 1 | 6
  Asian | 5 | 4 | 9
  Other | 7 | 2 | 9
MADRS Total Score [Mean (Standard Deviation); unit: score on a scale] — The MADRS is used to assess depressive symptom severity. It consists of 10 items (apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts and suicidal thoughts), each rated from 0 to 6 with zero being the "best" rating and 6 being the "worst" rating. The MADRS total score is the sum of ratings for all 10 items. The total score ranges from 0 to 60. A higher score on the MADRS represents a more severe level of depression. Population: Number analyzed is the number of participants with data available for analysis at the specified timepoint.
  score on a scale
    number analyzed (Participants) | 189 | 186 | 375
    (all) | 28.4 (6.0) | 28.4 (6.0) | 28.4 (6.0)
Generalized Anxiety Disorder-7 (GAD-7) Total Score [Mean (Standard Deviation); unit: score on a scale] — The GAD-7 is self-reported questionnaire designed to assess anxiety in participants. The scale contains 7 items (anxiety symptoms) and each item was rated by the participants from 0 (not at all) to 3 (nearly every day) based on how much they were bothered by each symptom. The total score ranges from 0 to 21. A higher score on the GAD-7 represents greater anxiety symptomatology. Population: Number analyzed is the number of participants with data available for analysis at the specified timepoint.
  score on a scale
    number analyzed (Participants) | 185 | 184 | 369
    (all) | 9.5 (4.5) | 9.7 (4.8) | 9.6 (4.7)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 6 in the MADRS Total Score
Description: The MADRS is used to assess depressive symptom severity. It consists of 10 items (apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts and suicidal thoughts), each rated from 0 to 6 with zero being the "best" rating and 6 being the "worst" rating. The MADRS total score is the sum of ratings for all 10 items. The total score ranges from 0 to 60. A higher score on the MADRS represents a more severe level of depression. A negative change from baseline indicates improvement. Least square (LS) mean was estimated using Mixed Model Repeated Measures (MMRM) method.
Time Frame: Baseline (Day 1) to Week 6
Population: FAS included all randomized participants who received at least 1 occurrence of either CT-152 or sham use and had baseline and at least 1 postbaseline assessment of MADRS total score. Overall number of participants analyzed is the number of participants with data available for analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Digital Therapeutic A - CT-152 | Digital Therapeutic B - Sham
Number analyzed (Participants) | 176 | 176
score on a scale | -9.03 (0.73) | -7.25 (0.73)
Statistical Analysis 1: Comparison: Digital Therapeutic A - CT-152 vs Digital Therapeutic B - Sham; Test type: Superiority; p = 0.0568, MMRM; p-value was calculated by MMRM method with model terms: Treatment, trial center, visit, treatment by visit, and baseline by visit interaction; Treatment Difference = -1.78, 95% CI 2-sided [-3.60 to 0.05]

2. Secondary Outcome: Change From Baseline to Week 6 in the GAD-7 Total Score
Description: The GAD-7 is self-reported questionnaire designed to assess anxiety in participants. The scale contains 7 items (anxiety symptoms) and each item was rated by the participants from 0 (not at all) to 3 (nearly every day) based on how much they were bothered by each symptom. The total score ranges from 0 to 21. A higher score on the GAD-7 represents greater anxiety symptomatology. A negative change from baseline indicates improvement. LS mean was estimated using MMRM method.
Time Frame: Baseline (Day 1) to Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Digital Therapeutic A - CT-152 | Digital Therapeutic B - Sham
Number analyzed (Participants) | 167 | 167
score on a scale | -3.41 (0.34) | -2.64 (0.34)
Statistical Analysis 1: Comparison: Digital Therapeutic A - CT-152 vs Digital Therapeutic B - Sham; Test type: Superiority; p = 0.0705, MMRM; [statistical method as in outcome 1, analysis 1]; Treatment Difference = -0.77, 95% CI 2-sided [-1.61 to 0.07]

3. Other Pre Specified Outcome: Change From Baseline to Weeks 2 and 4 in the MADRS Total Score
Description: The MADRS is used to assess depressive symptom severity. It consists of 10 items (apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts and suicidal thoughts), each rated from 0 to 6 with zero being the "best" rating and 6 being the "worst" rating. The MADRS total score is the sum of ratings for all 10 items. The total score ranges from 0 to 60. A higher score on the MADRS represents a more severe level of depression. A negative change from baseline indicates improvement. LS mean was estimated using MMRM method.
Time Frame: Baseline (Day 1) to Weeks 2 and 4
Population: FAS included all randomized participants who received at least 1 occurrence of either CT-152 or sham use and had baseline and at least 1 postbaseline assessment of MADRS total score. Overall number of participants analyzed is the number of participants with data available for analysis. Number analyzed is the number of participants with data available for analysis at the specified timepoints.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Digital Therapeutic A - CT-152 | Digital Therapeutic B - Sham
Number analyzed (Participants) | 176 | 176
score on a scale
  Week 2: number analyzed (Participants) | 175 | 171
  Week 2 | -3.85 (0.58) | -3.23 (0.59)
  Week 4: number analyzed (Participants) | 165 | 166
  Week 4 | -6.62 (0.67) | -5.16 (0.67)
Statistical Analysis 1: Comparison: Digital Therapeutic A - CT-152 vs Digital Therapeutic B - Sham; Week 2; Test type: Superiority; p = 0.3687, MMRM — p-value was calculated by MMRM method with model terms: Treatment, trial center, visit, treatment by visit, and baseline by visit interaction; Treatment Difference = -0.62, 95% CI 2-sided [-1.99 to 0.74]
Statistical Analysis 2: Comparison: Digital Therapeutic A - CT-152 vs Digital Therapeutic B - Sham; Week 4; Test type: Superiority; p = 0.0828, MMRM — [p-value comment as in outcome 3, analysis 1]; Treatment Difference = -1.45, 95% CI 2-sided [-3.10 to 0.19]

4. Other Pre Specified Outcome: Change From Baseline to Weeks 2 and 4 in the GAD-7 Total Score
Description: as for outcome 2
Time Frame: Baseline (Day 1) to Weeks 2 and 4
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Digital Therapeutic A - CT-152 | Digital Therapeutic B - Sham
Number analyzed (Participants) | 167 | 167
score on a scale
  Week 2: number analyzed (Participants) | 161 | 161
  Week 2 | -1.22 (0.30) | -0.88 (0.30)
  Week 4: number analyzed (Participants) | 157 | 153
  Week 4 | -2.22 (0.33) | -1.93 (0.33)
Statistical Analysis 1: Comparison: Digital Therapeutic A - CT-152 vs Digital Therapeutic B - Sham; Week 2; Test type: Superiority; p = 0.3549, MMRM — [p-value comment as in outcome 3, analysis 1]; Treatment Difference = -0.34, 95% CI 2-sided [-1.06 to 0.38]
Statistical Analysis 2: Comparison: Digital Therapeutic A - CT-152 vs Digital Therapeutic B - Sham; Week 4; Test type: Superiority; p = 0.4948, MMRM — [p-value comment as in outcome 3, analysis 1]; Treatment Difference = -0.28, 95% CI 2-sided [-1.09 to 0.53]

5. Other Pre Specified Outcome: MADRS Response Rate at Weeks 2, 4, and 6
Description: The MADRS is used to assess depressive symptom severity. It consists of 10 items (apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts and suicidal thoughts), each rated from 0 to 6 with zero being the "best" rating and 6 being the "worst" rating. The MADRS total score is the sum of ratings for all 10 items. The total score ranges from 0 to 60. A higher score on the MADRS represents a more severe level of depression. MADRS Response Rate was defined as the percentage of participants who achieved a reduction in the MADRS total score by 50% or more from baseline.
Time Frame: Baseline (Day 1), Weeks 2, 4 and 6
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Digital Therapeutic A - CT-152 | Digital Therapeutic B - Sham
Number analyzed (Participants) | 176 | 176
percentage of participants
  Week 2: number analyzed (Participants) | 175 | 171
  Week 2 | 10.86 | 5.85
  Week 4 | 18.18 | 13.64
  Week 6 | 28.41 | 20.45
Statistical Analysis 1: Comparison: Digital Therapeutic A - CT-152 vs Digital Therapeutic B - Sham; Week 2; Test type: Superiority; p = 0.1420, Cochran-Mantel-Haenszel — p-value was calculated by Cochran-Mantel-Haenzsel general association test controlling for study center; Ratio of Response Rate = 1.68, 95% CI 2-sided [0.84 to 3.34]
Statistical Analysis 2: Comparison: Digital Therapeutic A - CT-152 vs Digital Therapeutic B - Sham; Week 4; Test type: Superiority; p = 0.2939, Cochran-Mantel-Haenszel — p-value was calculated by Cochran-Mantel-Haenzsel general association test controlling for study center; Ratio of Response Rate = 1.31, 95% CI 2-sided [0.79 to 2.16]
Statistical Analysis 3: Comparison: Digital Therapeutic A - CT-152 vs Digital Therapeutic B - Sham; Week 6; Test type: Superiority; p = 0.0884, Cochran-Mantel-Haenszel — p-value was calculated by Cochran-Mantel-Haenzsel general association test controlling for study center; Ratio of Response Rate = 1.38, 95% CI 2-sided [0.96 to 1.99]

6. Other Pre Specified Outcome: Change From Baseline to Weeks 2, 4 and 6 in the Clinical Global Impression - Severity of Illness (CGI-S) Score
Description: The CGI-S is a standardized, clinician-administered global rating scale that measures disease severity on a 7-point Likert scale To perform this assessment, the investigator (or designee) answered the following question: "Considering your total clinical experience with this particular population, how mentally ill (as related to agitation) is the participant at this time?" Response choices are 0 = not assessed; 1 = normal, not at all ill; 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; and 7 = among the most extremely ill subjects. The score 0 (not assessed) will be set to missing. LS mean was estimated using MMRM method.
Time Frame: Baseline (Day 1) to Weeks 2, 4 and 6
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Digital Therapeutic A - CT-152 | Digital Therapeutic B - Sham
Number analyzed (Participants) | 175 | 172
score on a scale
  Week 2 | -0.54 (0.06) | -0.34 (0.06)
  Week 4: number analyzed (Participants) | 166 | 166
  Week 4 | -0.84 (0.07) | -0.52 (0.07)
  Week 6: number analyzed (Participants) | 160 | 155
  Week 6 | -1.06 (0.08) | -0.80 (0.08)
Statistical Analysis 1: Comparison: Digital Therapeutic A - CT-152 vs Digital Therapeutic B - Sham; Week 2; Test type: Superiority; p = 0.0039, MMRM — [p-value comment as in outcome 3, analysis 1]; Treatment Difference = -0.19, 95% CI 2-sided [-0.32 to -0.06]
Statistical Analysis 2: Comparison: Digital Therapeutic A - CT-152 vs Digital Therapeutic B - Sham; Week 4; Test type: Superiority; p = 0.0003, MMRM — [p-value comment as in outcome 3, analysis 1]; Treatment Difference = -0.32, 95% CI 2-sided [-0.50 to -0.15]
Statistical Analysis 3: Comparison: Digital Therapeutic A - CT-152 vs Digital Therapeutic B - Sham; Week 6; Test type: Superiority; p = 0.0098, MMRM — [p-value comment as in outcome 3, analysis 1]; Treatment Difference = -0.26, 95% CI 2-sided [-0.46 to -0.06]

7. Other Pre Specified Outcome: Change From Baseline to Week 6 in the World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0) Total Score
Description: The WHODAS 2.0 is a 36-item self-assessment scale to measure a participant's function and disability across 6 domains of life: cognition (understanding & communicating), mobility (moving & getting around), self-care (hygiene, dressing, eating, staying alone), getting along (interacting with others), life activities (domestic responsibilities, leisure, work & school), & participation (community & society). Each item is rated from 0 (none) to 4 (extreme or cannot do). The total score of the 36 items is converted into a metric ranging from 0 (no-disability) to 100 (full- disability) by dividing the total score by the maximum possible value of the total score, which is 144 for 36 items and multiplying by 100. LS Mean was estimated using ANCOVA method.
Time Frame: Baseline (Day 1) to Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Digital Therapeutic A - CT-152 | Digital Therapeutic B - Sham
Number analyzed (Participants) | 157 | 155
score on a scale | -5.58 (1.15) | -4.56 (1.18)
Statistical Analysis 1: Comparison: Digital Therapeutic A - CT-152 vs Digital Therapeutic B - Sham; Test type: Superiority; p = 0.4463, ANCOVA — p-value was calculated by ANCOVA model, with treatment and study center as main effects and baseline value as covariate; Treatment Difference = -1.02, 95% CI 2-sided [-3.66 to 1.61]

8. Other Pre Specified Outcome: Change From Screening to Weeks 4 and 6 in the PHQ-9 Total Score.
Description: The PHQ-9 is a standardized, self-administered rating scale that assesses the severity of depressive symptoms. The scale consists of 9 items, representing the 9 criteria upon which the diagnosis of DSM-IV depressive disorders is based. Each item is rated from 0 (not at all) to 3 (nearly every day). The total score ranges from 0 to 27. A higher score on the PHQ-9 represents a higher severity of depressive symptoms. LS mean was estimated using MMRM method.
Time Frame: Screening to Weeks 4 and 6
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Digital Therapeutic A - CT-152 | Digital Therapeutic B - Sham
Number analyzed (Participants) | 160 | 157
score on a scale
  Week 4 | -5.14 (0.43) | -3.85 (0.45)
  Week 6: number analyzed (Participants) | 153 | 152
  Week 6 | -6.68 (0.45) | -5.10 (0.46)
Statistical Analysis 1: Comparison: Digital Therapeutic A - CT-152 vs Digital Therapeutic B - Sham; Week 4; Test type: Superiority; p = 0.0102, MMRM — [p-value comment as in outcome 3, analysis 1]; Treatment Difference = -1.29, 95% CI 2-sided [-2.28 to -0.31]
Statistical Analysis 2: Comparison: Digital Therapeutic A - CT-152 vs Digital Therapeutic B - Sham; Week 6; Test type: Superiority; p = 0.0029, MMRM — [p-value comment as in outcome 3, analysis 1]; Treatment Difference = -1.58, 95% CI 2-sided [-2.62 to -0.54]

9. Other Pre Specified Outcome: MADRS Partial Response at Weeks 2, 4 and 6
Description: The MADRS is used to assess depressive symptom severity. It consists of 10 items (apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts and suicidal thoughts), each rated from 0 to 6 with zero being the "best" rating and 6 being the "worst" rating. The MADRS total score is the sum of ratings for all 10 items. The total score ranges from 0 to 60. A higher score on the MADRS represents a more severe level of depression. MADRS partial response was defined as the percentage of participants who achieved a reduction in the MADRS total score by 30% or more and less than 50% from baseline.
Time Frame: Baseline (Day 1), Weeks 2, 4 and 6
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Digital Therapeutic A - CT-152 | Digital Therapeutic B - Sham
Number analyzed (Participants) | 176 | 176
percentage of participants
  Week 2: number analyzed (Participants) | 175 | 171
  Week 2 | 13.14 | 11.11
  Week 4 | 19.32 | 16.48
  Week 6 | 19.89 | 17.05
Statistical Analysis 1: Comparison: Digital Therapeutic A - CT-152 vs Digital Therapeutic B - Sham; Week 2; Test type: Superiority; p = 0.5757, Cochran-Mantel-Haenszel — p-value was calculated by Cochran-Mantel-Haenzsel general association test controlling for study center; Ratio of Response Rate = 1.18, 95% CI 2-sided [0.65 to 2.16]
Statistical Analysis 2: Comparison: Digital Therapeutic A - CT-152 vs Digital Therapeutic B - Sham; Week 4; Test type: Superiority; p = 0.5102, Cochran-Mantel-Haenszel — p-value was calculated by Cochran-Mantel-Haenzsel general association test controlling for study center; Ratio of Response Rate = 1.16, 95% CI 2-sided [0.75 to 1.78]
Statistical Analysis 3: Comparison: Digital Therapeutic A - CT-152 vs Digital Therapeutic B - Sham; Week 6; Test type: Superiority; p = 0.5342, Cochran-Mantel-Haenszel — p-value was calculated by Cochran-Mantel-Haenzsel general association test controlling for study center; Ratio of Response Rate = 1.15, 95% CI 2-sided [0.74 to 1.79]

10. Other Pre Specified Outcome: MADRS Response Rate at Weeks 8 and 10
Description: The MADRS is used to assess depressive symptom severity. It consists of 10 items (apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts and suicidal thoughts), each rated from 0 to 6 with zero being the "best" rating and 6 being the "worst" rating. The MADRS total score is the sum of ratings for all 10 items. The total score ranges from 0 to 60. A higher score on the MADRS represents a more severe level of depression. MADRS Response Rate (full or partial) was defined as the percentage of participants who achieved a reduction in the MADRS total score by 30% or more from baseline.
Time Frame: Baseline (Day 1), Weeks 8 and 10
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Digital Therapeutic A - CT-152 | Digital Therapeutic B - Sham
Number analyzed (Participants) | 168 | 160
percentage of participants
  Week 8: number analyzed (Participants) | 164 | 155
  Week 8 | 54.88 | 54.84
  Week 10 | 60.71 | 57.50
Statistical Analysis 1: Comparison: Digital Therapeutic A - CT-152 vs Digital Therapeutic B - Sham; Week 8; Test type: Superiority; Ratio of Response Rate = 1.00, 95% CI 2-sided [0.82 to 1.22]
Statistical Analysis 2: Comparison: Digital Therapeutic A - CT-152 vs Digital Therapeutic B - Sham; Week 10; Test type: Superiority; Ratio of Response Rate = 1.05, 95% CI 2-sided [0.88 to 1.25]

ADVERSE EVENTS:
Time Frame: From the signing of the informed consent up to end of study (up to Week 10)
Description: Safety sample included all randomized participants who received at least 1 occurrence of either CT-152 or sham use.
Arm/Group | Digital Therapeutic A - CT-152 | Digital Therapeutic B - Sham
All-Cause Mortality (participants affected / at risk) | 0/187 | 0/186
Serious Adverse Events (participants affected / at risk) | 1/187 | 0/186
Other Adverse Events (participants affected / at risk) | 3/187 | 10/186
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Digital Therapeutic A - CT-152 (N=187) | Digital Therapeutic B - Sham (N=186)
Transient Ischaemic Attack (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Digital Therapeutic A - CT-152 (N=187) | Digital Therapeutic B - Sham (N=186)
Upper Respiratory Tract Infection (Infections and infestations) | 3 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-11-03): https://cdn.clinicaltrials.gov/large-docs/85/NCT04770285/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-16): https://cdn.clinicaltrials.gov/large-docs/85/NCT04770285/SAP_001.pdf